CLINICAL TRIAL: NCT02068508
Title: Actos Tablets Special Drug Use Surveillance "Combined Use of Insulin Products / Long-term Treatment"
Brief Title: Pioglitazone Tablets Special Drug Use Surveillance "Combined Use of Insulin Products / Long-term Treatment"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 237-018; JapicCTI-132376 (Registry Identifier: JapicCTI); JapicCTI-R171012 (Other: JapicCTI)
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pioglitazone: Pioglitazone 15 mg to 30 mg, orally, once daily
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone Tablets
  Other Names: Actos

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of long-term treatment with pioglitazone (Actos Tablets) in the routine clinical setting in combination with an insulin product in patients with type 2 diabetes mellitus who responded inadequately when using an insulin product in addition to diet therapy and exercise therapy.

DETAILED DESCRIPTION:
This is a special drug use surveillance on long-term use of newly co-administered pioglitazone tablets (Actos Tablets) as part of routine medical care in patients with type 2 diabetes mellitus who have poorly controlled blood glucose when using an insulin product in addition to diet therapy and exercise therapy; this survey is designed to determine the safety and efficacy of long-term use of pioglitazone tablets (Actos Tablets) in the routine clinical setting in combination with an insulin product (the planned sample size, 1000.) The usual adult dosage is 15 mg of pioglitazone administered orally once daily before or after breakfast. Dose adjustment will be made according to gender, age, and symptoms with an upper limit of 30 mg.

ELIGIBILITY:
Inclusion Criteria:

Participants with type 2 diabetes mellitus assumed to have insulin resistance who responded inadequately when using an insulin product in addition to diet therapy and exercise therapy who meet the following criteria at enrollment.

1. Participants treated with an insulin product for at least 4 weeks
2. Participants who started Actos Tablets for the first time after the start of an insulin product
3. Participants likely to be available for a 52-week observation and evaluation after the start of co-administration of Actos Tablets

Exclusion Criteria:

Participants with contraindications to Actos Tables and insulin products treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 1067 (Actual)
Dates: Start 2009-07-30 (Actual); Primary Completion 2014-06-30 (Actual); Study Completion 2014-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: No
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 169 investigative sites in Japan, from 30-July-2009 to 30-June-2014.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus who failed to respond adequately to treatment with insulin therapy were enrolled to receive pioglitazone 15 milligram (mg) - 30 mg for up to 12 months. Participants received interventions as part of routine medical care.
Groups:
- Pioglitazone: Pioglitazone 15 mg - 30 mg, tablet, orally, once daily for up to 12 months in participants based upon the disease severity. Participants will receive interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Pioglitazone
Started | 1067
Completed | 1035
Not Completed | 32
Not completed — Case report forms uncollected | 27
Not completed — Patient did not visit the study site | 1
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1035
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (12.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 477
  Male | 558
Region of Enrollment [Number; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 1035
Pregnancy Status [Count of Participants; unit: Participants] — This baseline characteristic was analyzed only in female participants.
  Participants
    Pregnant | 0
    Not pregnant | 477
Duration of type 2 diabetes mellitus [Count of Participants; unit: Participants] — Mean Duration between start of study and first time of diagnosis of type 2 diabetes mellitus was reported.
  Participants
    < 1 year | 27
    ≥ 1 year < 5 years | 98
    ≥ 5 years < 10 years | 199
    ≥ 10 years | 661
    Unknown | 50
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had Predisposition to Hypersensitivity | 48
    Had No Predisposition to Hypersensitivity | 983
    Unknown | 4
Drinking Habits [Count of Participants; unit: Participants]
  Never Drank | 661
  Ex-Drinker | 77
  Current Drinker | 280
  Unknown | 17
Smoking Habits [Count of Participants; unit: Participants]
  Never Smoked | 687
  Ex-Smoker | 160
  Current Smoker | 162
  Unknown | 26
Body Weight [Mean (Standard Deviation); unit: kg] | 65.849 (14.0584)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 25.45 (4.336)
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above. Participants may be represented in more than 1 category.
  Participants
    Had Presence of Medical History | 343
    Had No Presence of Medical History | 683
    Unknown | 9
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above. Participants may be represented in more than 1 category.
  Participants
    Had Presence of Medical Complications | 957
    Had Presence of Medical No Complications | 78
Concomitant Hepatic Disease [Count of Participants; unit: Participants]
  Had Concomitant Hepatic Disease | 126
  Had No Concomitant Hepatic Disease | 909
Concomitant Renal Disease [Count of Participants; unit: Participants]
  Had Concomitant Renal Disease | 423
  Had No Concomitant Renal Disease | 612
Concomitant Cardiac Disease [Count of Participants; unit: Participants]
  Had Concomitant Cardiac Disease | 148
  Had No Concomitant Cardiac Disease | 887
Diabetic Complications [Count of Participants; unit: Participants] — Number of Participants with Any of Diabetic Retinopathy, Diabetic Nephropathy, and Diabetic Neuropathy at Start of Study Treatment was reported.
  Participants
    Had Diabetic Complications | 633
    Had No Diabetic Complications | 402
Diet Therapy [Count of Participants; unit: Participants]
  On Diet Therapy | 1000
  Not on Diet Therapy | 34
  Unknown | 1
Exercise Therapy [Count of Participants; unit: Participants]
  On Exercise Therapy | 932
  Not on Exercise Therapy | 102
  Unknown | 1
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dL] | 172.0 (65.49)
Haemoglobin A1c (HbA1c) [National Glycohemoglobin Standardization Program (NGSP)] [Mean (Standard Deviation); unit: Percent] | 8.72 (1.449)
Fasting Triglyceride [Mean (Standard Deviation); unit: mg/dL] | 156.5 (133.21)
HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 55.92 (17.205)
LDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 111.46 (28.418)
Serum creatinine (Enzymatic method) [Mean (Standard Deviation); unit: mg/dL] | 0.784 (0.2853)
Urine protein (Qualitative) [Count of Participants; unit: Participants] — Data of urine protein tests were reported, The test detect and/or measure protein being released into the urine. The stages of reported data were "- = absent", "± = 15 mg/dL", "+ = 30 mg/dL", "2+ = 100 mg/dL", "3+ = 300 mg/dL" respectively.
  Participants
    - | 501
    ± | 140
    ＋ | 101
    2＋ | 66
    3＋ | 30
    Unknown/No measuremen | 197
Urine albumin/Creatinine ratio [Mean (Standard Deviation); unit: mg/gCR] | 169.616 (535.5513)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 131.6 (15.17)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 73.7 (10.53)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Adverse Drug Reactions (ADRs)
Description: ADRs are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Up to Week 52
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1035
Participants | 213

2. Secondary Outcome: Change From Baseline in Fasting Blood Glucose
Time Frame: Baseline and Week 12, 24, 36, 52, and final assessment (up to Week 52)
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available. Here number of participants analyzed was evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1013
mg/dL
  Change at Week 12: number analyzed (Participants) | 441
  Change at Week 12 | -26.2 (60.97)
  Change at Week 24: number analyzed (Participants) | 390
  Change at Week 24 | -23.9 (60.55)
  Change at Week 36: number analyzed (Participants) | 326
  Change at Week 36 | -21.7 (64.72)
  Change at Week 52: number analyzed (Participants) | 336
  Change at Week 52 | -21.4 (65.47)
  Change at Final Assessment: number analyzed (Participants) | 500
  Change at Final Assessment | -23.8 (69.96)

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Time Frame: Baseline and Week 12, 24, 36, 52, and final assessment (up to Week 52)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1013
Percent
  Change at Week 12: number analyzed (Participants) | 880
  Change at Week 12 | -0.62 (1.024)
  Change at Week 24: number analyzed (Participants) | 754
  Change at Week 24 | -0.75 (1.210)
  Change at Week 36: number analyzed (Participants) | 696
  Change at Week 36 | -0.77 (1.192)
  Change at Week 52: number analyzed (Participants) | 661
  Change at Week 52 | -0.75 (1.169)
  Change at Final Assessment: number analyzed (Participants) | 927
  Change at Final Assessment | -0.72 (1.236)

4. Secondary Outcome: Change From Baseline in Fasting Triglycerides
Time Frame: Baseline and Week 12, 24, 36, 52, and final assessment (up to Week 52)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1013
mg/dL
  Change at Week 12: number analyzed (Participants) | 438
  Change at Week 12 | -20.7 (90.24)
  Change at Week 24: number analyzed (Participants) | 395
  Change at Week 24 | -19.8 (109.61)
  Change at Week 36: number analyzed (Participants) | 339
  Change at Week 36 | -28.4 (123.98)
  Change at Week 52: number analyzed (Participants) | 340
  Change at Week 52 | -8.5 (115.86)
  Change at Final Assessment: number analyzed (Participants) | 503
  Change at Final Assessment | -16.6 (128.17)

5. Secondary Outcome: Change From Baseline in HDL Cholesterol
Time Frame: Baseline and Week 12, 24, 36, 52, and final assessment (up to Week 52)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1013
mg/dL
  Change at Week 12: number analyzed (Participants) | 671
  Change at Week 12 | 3.32 (8.898)
  Change at Week 24: number analyzed (Participants) | 598
  Change at Week 24 | 1.98 (9.628)
  Change at Week 36: number analyzed (Participants) | 525
  Change at Week 36 | 1.79 (9.868)
  Change at Week 52: number analyzed (Participants) | 511
  Change at Week 52 | 1.35 (8.940)
  Change at Final Assessment: number analyzed (Participants) | 749
  Change at Final Assessment | 2.04 (9.358)

6. Secondary Outcome: Change From Baseline in LDL Cholesterol
Time Frame: Baseline and Week 12, 24, 36, 52, and final assessment (up to Week 52)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1013
mg/dL
  Change at Week 12: number analyzed (Participants) | 631
  Change at Week 12 | -0.96 (22.788)
  Change at Week 24: number analyzed (Participants) | 561
  Change at Week 24 | -0.16 (24.239)
  Change at Week 36: number analyzed (Participants) | 489
  Change at Week 36 | -0.68 (26.594)
  Change at Week 52: number analyzed (Participants) | 482
  Change at Week 52 | -0.33 (25.258)
  Change at Final Assessment: number analyzed (Participants) | 713
  Change at Final Assessment | -0.82 (25.908)

7. Secondary Outcome: Number of Participants Who Received Specific Daily Dose of Insulin Product at Each Time Points
Description: Number of participants who received study drug and specific daily dose of insulin product during the survey was reported. Daily dose of insulin was categorized by < 30 units, >= 30 and < 60 units, >= 60 and < 90 units, >= 90 units at each time points.
Time Frame: Baseline, Week 52, and final assessment (up to Week 52)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone
Number analyzed (Participants) | 1013
Participants
  Baseline: number analyzed (Participants) | 953
  Baseline: < 30 units of insulin product | 510
  Baseline: >= 30 and < 60 units of insulin product | 359
  Baseline: >= 60 and < 90 units of insulin product | 68
  Baseline: >= 90 units of insulin product | 16
  Week 52: number analyzed (Participants) | 697
  Week 52: < 30 units of insulin product | 379
  Week 52: >= 30 and < 60 units of insulin product | 256
  Week 52: >= 60 and < 90 units of insulin product | 52
  Week 52: >= 90 units of insulin product | 10
  Final Assessment: number analyzed (Participants) | 982
  Final Assessment: < 30 units of insulin product | 532
  Final Assessment: >= 30 and < 60 units of insulin product | 363
  Final Assessment: >= 60 and < 90 units of insulin product | 72
  Final Assessment: >= 90 units of insulin product | 15

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: At each visit the investigator had to document any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only ADRs were collected in this study. Participants may be represented in more than 1 category.
Arm/Group | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 11/1035
Other Adverse Events (participants affected / at risk) | 303/1035
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=1035)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Generalised oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone (N=1035)
Hypoglycaemia (Metabolism and nutrition disorders) | 163
Face oedema (General disorders) | 22
Oedema peripheral (General disorders) | 104
Weight increased (Investigations) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.